CLINICAL TRIAL: NCT04581668
Title: Impact of NAVA Ventilation on Brain Oxygenation and Perfusion in Children With Congenital Heart Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Dr Guillaume Emeriaud, Clinical Professor, St. Justine's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2021-2731
Record Dates: First submitted 2020-09-27; First posted 2020-10-09 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Tetralogy of Fallot; Hypoplastic Left Heart Syndrome; Univentricular Heart; Heart Defects, Congenital
MeSH Terms: conditions — Tetralogy of Fallot; Hypoplastic Left Heart Syndrome; Univentricular Heart; Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Cross over physiological study with 2 different phases with a 30 minute Wash out period: 30 minutes. Order will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurally adjusted ventilatory assist first (Other): Ventilation in NAVA mode then ventilation in conventional mode
  Interventions: Other: Neurally adjusted ventilatory assist first
- Conventional ventilation first (Other): Ventilation in conventional mode then ventilation in NAVA mode
  Interventions: Other: Conventional ventilation first

INTERVENTIONS:
Other: Neurally adjusted ventilatory assist first — Invasive ventilation in Neurally adjusted ventilatory assist during 60 minutes followed by a 30 minutes wash out period then ventilation in conventional mode
  Arms: Neurally adjusted ventilatory assist first
Other: Conventional ventilation first — Invasive ventilation in conventional mode during 60 minutes followed by a 30 minutes wash out period then ventilation in Neurally adjusted ventilatory assist
  Arms: Conventional ventilation first

SUMMARY:
Positive intra-thoracic pressures induced by mechanical ventilation can negatively impact right heart hemodynamics by restricting systemic venous return and increasing right ventricular afterload. These consequences may be detrimental in patients with a restrictive right ventricular physiology and in patients with single ventricle physiology. NAVA (Neurally Adjusted Ventilatory Assist) ventilation decreases intra thoracic pressures compared to conventional ventilation modes. Brain perfusion is both a hemodynamic indicator and a prognostic factor in cardiac postoperative care. Diffuse Correlation Spectroscopy (DCS) coupled with Near Infrared Spectroscopy (NIRS) is a new technology that allows monitoring, in addition to brain tissue oxygenation, changes in brain blood flow.

This physiological study aims to evaluate the impact of NAVA mode ventilation on cerebral and systemic hemodynamics in post-operative cardiac surgery patients with preload dependant right ventricle or with passive venous return to the lungs . This prospective cross-over study will include 30 patients.

Once stabilized in intensive care, patients will undergo 2 periods of ventilation in NAVA mode and conventional mode separated by a 30-minute washout period, in a random order.

For each period the following information will be collected: changes in cerebral blood flow and cerebral oxygenation, hemodynamic parameters including cardiac output and oxygen transport and ventilatory parameters.

DETAILED DESCRIPTION:
1. Scientific context

   In post-operative cardiac surgery, invasive ventilation is often necessary, but the induced positive intra thoracic pressures can be detrimental to hemodynamics via several mechanisms: decrease in venous return, increase in pulmonary vascular resistance and increase in the afterload of the right ventricle. This effect is particularly problematic in patients with a restrictive right ventricle, who are preload dependent, and in patients with cavo pulmonary connections for single ventricle palliation. In these patients, decreasing ventilator positive pressure improves cardiac output and cerebral oxygenation. However, very early extubation is not always possible or safe, and it is therefore essential to optimize mechanical ventilation in order to minimize its hemodynamic consequences.

   In adults, ventilation in NAVA (Neurally Adjusted Ventilatory Assist) mode, regardless of the level of assistance, allows the preservation of intra thoracic pressure variations characteristic of spontaneous ventilation and limits the impact of ventilation on right ventricular ejection. In children, inspiratory and mean pressures are also lower in NAVA compared to conventional ventilation.

   Assessment of brain oxygenation and perfusion in cardiovascular resuscitation is important both as a hemodynamic parameter and as a neurological prognostic factor. An innovative non-invasive tool, Diffuse Correlation Spectroscopy coupled with Near Infrared Spectroscopy (DCS-NIRS), allows the non-invasive evaluation of both cerebral oxygenation and variations in cerebral blood flow.
2. Hypothesis and objectives

   The hypothesis is that the NAVA ventilation mode, which generates lower intra thoracic pressures than conventional ventilation modes, will improve cerebral hemodynamics, cardiac output, and oxygen transport of at-risk patients in the post-operative cardiac surgery setting compared with conventional ventilation.

   Main objective:

   In pediatric patients following cardiac surgery with risk of right ventricular diastolic dysfunction or passive pulmonary venous return (including Glenn, hemi-Fontan, Fontan, and Tetralogy of Fallot surgery), investigators will evaluate the impact of NAVA ventilation on:
   * cerebral perfusion: cerebral blood flow (mm2/s) measured by DCS.
   * cerebral oxygenation: cerebral tissue saturation (%) and regional cerebral O2 extraction (OEF, measured by NIRS-DCS).

   Secondary objective:

   In pediatric post-operative cardiac surgery patients with risk of restrictive right ventricle or passive pulmonary venous return (including Glenn, hemi-Fontan, Fontan, and Tetralogy of Fallot type surgery), investigators will compare the impact of conventional ventilation to NAVA mode on:
   * Brain regional O2 consumption extracted from NIRS-DCS measurements
   * Systemic hemodynamics, including cardiac index, lactate level, central venous oxygen saturation (ScvO2), and oxygen transport
   * Ventilation parameters
   * Comfort as measured by the COMFORT scale
3. Methods

This is a prospective cross-over, single-center, physiological study to be conducted in the Pediatric Intensive Care Unit of CHU Sainte Justine (Montreal, Canada).

Two periods of 60 minutes in each of 2 ventilation modes will be compared: conventional ventilation mode (as prescribed by the treating team) and NAVA mode, in random order.

On admission to the PICU postoperatively, study patients will be fitted with a naso-gastric NAVA probe.

Before performing any study measurements, investigators will wait for patient stabilization, which is defined by:

* absence of hemodynamically significant bleeding
* stabilization of the ventilation parameters
* stable inotrope dose The order of the 2 ventilation periods will be randomized according to a previously generated random list.

Study period ventilation will be set as follows:

* conventional ventilation: ventilation as prescribed by the treating team will be continued. Usually, ventilation is in PRVC (pressure regulated volume control) mode with a tidal volume between 5 and 8 mL/kg, a peep between 4 and 5, a respiratory rate to aim for normocapnia, and FiO2 to aim for PaO2 between 100 and 150 mmHg.
* NAVA Mode: NAVA level setting to target an Edi level between 3 and 20 V, tidal volume between 5 and 7 mL/kg, and no respiratory distress on physical examination. The trigger will be set at 0.5 V. The maximum pressure will be limited to 30 cmH2O. The PEEP level will not be changed from that prescribed by the treating physician.

To facilitate comparability of brain flow and oxygenation measurements, FiO2, NO concentration, inotrope dose, and sedation will be kept as stable as possible during these periods, at the discretion of the treating physician. Similarly, if possible, blood transfusions will not be administered during the study period.

During the two periods of ventilation, the following parameters will be recorded continuously:

* ventilatory parameters: ventilator parameters according to the set mode: peak inspiratory pressure, mean airway pressure, PEEP, tidal volume, total and spontaneous minute ventilation, Edi level, FiO2, exhaled CO2 via volumetric capnography.
* hemodynamic parameters: heart rate (HR), mean arterial pressure, systolic, diastolic, central venous pressure (CVP), left atrial pressure (LAP), type and dose of vasoactive medications received with calculation of the vasoactive-inotropic score.

In the second half of each period, investigators will perform:

* a central arterial and venous blood gas and an arterial lactate measurement.
* a measurement of cerebral blood flow by diffuse correlation spectroscopy and a measurement of cerebral regional tissue saturation and oxygen extraction. These measurements are done non-invasively and painlessly by applying a probe to the child's forehead for approximately 20 minutes.
* a limited cardiac ultrasound for the calculation of cardiac output (CO).
* calculation of urine output during the ventilation period.

In addition, for each patient, the following information will be collected:

* age at the time of surgery
* cardiac diagnosis
* existence and quantification of aorto-pulmonary collaterals
* preoperative medications
* operative details: surgical procedure, duration of cardiopulmonary bypass, aortic cross-clamp duration, inotropes administered (and maximum dose).
* result of the postoperative trans-esophageal cardiac echo (cardiac function, evaluation of repair, presence of residual anatomic lesions)
* arterial and venous blood gases, lactate and haemoglobin levels prior to study ventilation periods
* time interval between the end of cardiopulmonary bypass and the start of study measurements

The variables will be expressed in terms of mean standard deviation or median (interquartile), depending on the nature of their distribution. Because of the sample size, analysis of the differences between t variables during the 2 modes of ventilation will be done using the non-parametric Wilcoxon test (all the variables studied are of the continuous type). A value of p <0.05 will be considered significant.

For the calculation of sample size, investigators estimated, using the study by Huang et al (4), that the standard deviation of brain saturation would be 6%, and that the expected difference between the 2 ventilation modes would be at least 6%. To reach a power of 90% with an alpha risk set at 0.05, a minimum of 24 patients is required. Given the risk of loss of sight (e.g. technical difficulty in obtaining the main variable) and due to the heterogeneity of the patient population, we decided to aim to include 30 patients.

Note that no power calculation based on the variations in cerebral blood flow measured in spectroscopy was performed, because there was no preliminary data on the subject.

Approval from the Research Ethics Committee of Sainte Justine University Hospital and the University Medical Affairs Department was obtained. Written consent will be required from the parents.

ELIGIBILITY:
Inclusion Criteria:

1. admission to the pediatric intensive care unit:

   * after Glenn, Fontan, Fallot Tetralogy surgery
   * or after other types of surgery with risk of post-operative occurence of right ventricular failure or low lung output
2. invasive ventilation scheduled for at least 2 hours after admission

Exclusion Criteria:

* Contraindication to placement of a nasogastric NAVA tube
* History of significant focal brain injury (infarction or hemorrhage)
* Bilateral phrenic paralysis
* Extubation in operating room or planned to be within the hour,
* Patient with open chest, uncontrolled shock, need for neuromuscular blockade. Note that for these criteria, the patient may become eligible when these criteria are resolved.
* Patients for whom an acute care limitation order is in place.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Brain perfusion | 30 minutes
  cerebral blood flow measured with diffuse correlation spectroscopy (mm2/s)
Brain oxygenation | 30 minutes
  cerebral tissue saturation measured with near-infrared spectroscopy (%)
Brain oxygen extraction | 30 minutes
  Cerebral tissue oxygen extraction measured with near-infrared spectroscopy (%)

SECONDARY OUTCOMES:
Brain regional oxygen consumption | 30 minutes
  Cerebral tissue oxygen extraction measured with near-infrared spectroscopy
Cardiac output | 30 minutes
  Cardiac output measured using sub aortic time-velocity integral measured on cardiac ultrasound
Cardiac index | 30 minutes
  Cardiac index measured using sub aortic time-velocity integral measured on cardiac ultrasound
Oxygen transport | 50 minutes
  According to the following calculation: 1.34 x hemoglobin x SaO2 + 0.0031 x PaO2
Mean airway pressure (cmH2O) | 60 minutes
  Mean airway pressure (cmH2O) extracted from the ventilator every 30 seconds
Tidal volume | 60 minutes
  extracted from the ventilator every 30 seconds
Respiratory rate | 60 minutes
  extracted from the ventilator every 30 seconds
Minute ventilation | 60 minutes
  extracted from the ventilator every 30 seconds
Electrical activity of the diaphragm | 60 minutes
  extracted from the ventilator every 30 seconds
PaO2/FiO2 ratio | 50 minutes
  Ratio calculated at the end of each ventilation period, based on arterial blood gas

OTHER OUTCOMES:
Patient comfort | 60 minutes
  Measured by the COMFORT-B scale (ranges: 6-30, the lowest being the better)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Emeriaud, Dr, Principal Investigator — St. Justine's Hospital
Locations (1):
- St. Justine's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided